CLINICAL TRIAL: NCT06539169
Title: FLOWER: Following Longitudinal Outcomes With Epidemiology for Rare Diseases
Status: Recruiting | Type: Observational
Sponsor: xCures (Industry)
Responsible Party: Sponsor
Other Study IDs: XC-FLW-2024
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-08

CONDITIONS: Alpha-Thalassemia; Beta-Thalassemia; Amyloidosis; Amyotrophic Lateral Sclerosis; Creutzfeld-Jakob Disease; Cystic Fibrosis; Duchenne Muscular Dystrophy; Early-Onset Alzheimer Disease; Ehlers-Danlos Syndrome; Huntington Disease; Gaucher Disease; GM1 Gangliosidosis; Myasthenia Gravis; Pompe Disease; Sickle Cell Disease; Transthyretin Amyloid Cardiomyopathy; Rare Diseases
Keywords: rare diseases
MeSH Terms: conditions — alpha-Thalassemia; beta-Thalassemia; Amyloidosis; Amyotrophic Lateral Sclerosis; Insomnia, Fatal Familial; Cystic Fibrosis; Muscular Dystrophy, Duchenne; Alzheimer Disease; Ehlers-Danlos Syndrome; Huntington Disease; Gaucher Disease; Gangliosidosis, GM1; Myasthenia Gravis; Glycogen Storage Disease Type II; Anemia, Sickle Cell; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
FLOWER is a completely virtual, nationwide, real-world observational study to collect, annotate, standardize, and report clinical data for rare diseases. Patients participate in the study by electronic consent (eConsent) and sign a medical records release to permit data collection. Medical records are accessed from institutions directly via eFax or paper fax, online from patient electronic medical record (EMR) portals, direct from DNA/RNA sequencing and molecular profiling vendors, and via electronic health information exchanges. Patients and their treating physicians may also optionally provide medical records. Medical records are received in or converted to electronic/digitized formats (CCDA, FHIR, PDF), sorted by medical record type (clinic visit, in-patient hospital, out-patient clinic, infusion and out-patient pharmacies, etc.) and made machine-readable to support data annotation, full text searches, and natural language processing (NLP) algorithms to further facilitate feature identification.

DETAILED DESCRIPTION:
This study does not require data entry by treating site staff or physicians. Centralized data structuring is completed by xCures study staff. Data elements are aggregated, normalized, and coded to OMOP-based ontologies (SNOMED, LOINC, ICD-10, CTCAE, RxNorm, and MedDRA) in one process, permitting standardization of verbatim terms from medical records. The data collection platform supports 21 CFR Part 11-compliant data annotation with formal QC/QA process, medical review, and source data verification.

Beyond EMR data, raw DICOM images (MRI, CT files) can be collected from all sites of care and anonymized for integration with the clinical data. Molecular profiling and somatic or germline genomics results, and biochemical lab data, when available, are collected from commercial and academic sources and centralized. Additionally, patient- and caregiver-reported outcome surveys (PROs) can be collected to supplement information not found in clinical records.

Together, these clinical, imaging, biomarker, and assessment data will provide a comprehensive and longitudinal documentation of rare diseases in near real-time in a single observational basket study.

Traditional rare disease research registries rely on patients reporting many aspects of their condition via surveys or rely on key opinion leaders at specific institutions managing a team to enroll patients and annotate necessary data. These put unnecessary burdens on patients and strain limited research resources at medical centers. Gathering the necessary data and in sufficient quantities is often a limitation to successfully defining the natural history of a rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Any person with a known or suspected rare disease, defined by their prevalence of fewer than 200,000 individuals nationwide. Diseases include but are not limited to:

Alpha- or Beta- Thalassemia Amyloidosis Amyotrophic Lateral Sclerosis (ALS) Creutzfeldt-Jakob disease (CJD) Cystic Fibrosis (CF) Duchenne Muscular Dystrophy (DMD) Early-onset Alzheimer's Disease Ehlers-Danlos Syndrome (EDS) Huntington's Disease (HD) Gaucher Disease GM1 Gangliosidosis Myasthenia Gravis Pompe Disease Sickle Cell Disease Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Transthyretin Amyloid Polyneuropathy (ATTR-PN)

- Patients or their legally-authorized representative must be willing and able to provide informed consent (and assent, if applicable). Deceased persons may participate via consent of their legally-authorized representative in accordance with applicable Federal and state laws

Exclusion Criteria:

* Patient or LAR is unable to provide informed consent.
* Patient resides in a country other than the United States and is unable to provide access to medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include adult and pediatric patients with known or suspected rare disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 Years
Safety/tolerability of medications | 5 years
Changes in normal development milestones | 5 years
Changes in functional status | 5 years
Changes in motor function | 5 years
Changes in symptoms or clinical status | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- xCures, Los Altos, California, United States